CLINICAL TRIAL: NCT07224958
Title: ROAM OA: Functional and Patient Reported Outcomes Wearing a Knee Brace for Unicompartmental OA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: Enovis (Unknown)
Responsible Party: Principal Investigator, Markus Wimmer, Principal Investigator, Grainger Director of the RUSH Arthritis and Orthopedics Institute, Rush University Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 23110204-IRB01
Record Dates: First submitted 2025-10-28; First posted 2025-11-05 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Knee Osteoarthritis
Keywords: knee brace; gait analysis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Randomized crossover assignment followed by a parallel continuation period. Participants will cross over between the ROAM OA brace and the comparator, then continue in a chosen brace for the remainder of the study.
Masking Description: No blinding; all participants and study team are aware of the assigned brace.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- ROAM OA brace (Experimental): Participants receive the ROAM OA Single Upright Knee Brace (Enovis) to wear daily for the study duration. The brace is designed to offload the medial compartment of the knee and improve pain and function.
  Interventions: Device: ROAM OA Single Upright Knee Brace
- Active Comparator: Unloader brace or standard of care (Active Comparator): Participants receive the Ossur Unloader One knee brace or no brace (standard of care) and will follow standard pain management and physical therapy guidelines. This group serves as an active comparator to the ROAM OA brace.
  Interventions: Device: Ossur Unloader One Knee Brace or Standard of Care

INTERVENTIONS:
Device: ROAM OA Single Upright Knee Brace — A commercially available single-upright knee brace designed to offload the medial compartment of the knee in patients with unicompartmental osteoarthritis; manufactured by Enovis. Participants will wear the brace daily for the duration of the study.
  Arms: ROAM OA brace
Device: Ossur Unloader One Knee Brace or Standard of Care — Participants will receive the Ossur Unloader One knee brace or no brace (standard of care) and will follow standard management and physical therapy guidelines. This group serves as the active comparator to the ROAM OA brace.
  Arms: Active Comparator: Unloader brace or standard of care

SUMMARY:
The aim of this study is to conduct a comparative evaluation of the ROAM OA Single Upright Brace and the Ossur Unloader One Knee Brace in subjects with medial compartment osteoarthritis. The focus is on comparing the immediate and short-term biomechanical effects of these braces on knee adduction moments and spatiotemporal gait parameters, as well as assessing the long-term efficacy of the ROAM OA brace in improving pain and functional outcomes for individuals with osteoarthritis.

DETAILED DESCRIPTION:
INTRODUCTION The Enovis ROAM OA outcomes study is a prospective, single-center, crossover study with a subsequent randomized control phase and extended follow-up gait analysis, intended to evaluate the efficacy of the ROAM OA knee brace in subjects with medial knee osteoarthritis (OA).

The purpose of this study is to conduct a comparative evaluation of the ROAM OA Single Upright Brace and the Ossur Unloader One Knee Brace in subjects with medial compartment OA. The focus is on comparing the immediate and short-term biomechanical effects of these braces on knee adduction moments and spatiotemporal gait parameters, as well as assessing the long-term efficacy of the ROAM OA brace in improving pain and functional outcomes for individuals with OA.

1.1 Background Osteoarthritis of the knee significantly impacts the quality of life and functional capacity of those affected. Globally, hundreds of millions of people live with OA, with the knee being the most frequently affected joint. This condition leads to symptoms such as pain, swelling, and stiffness, which impair mobility and daily activities, affecting overall well-being and social connectedness.

The prevalence of knee OA is influenced by factors such as aging and obesity, and with an aging population, the incidence of knee OA is expected to rise. This increase underscores the need for effective management strategies.

Non-invasive interventions such as knee orthoses have been highlighted in OA management. These devices, including the ROAM OA Single Upright Brace, are designed to unload the affected compartment of the knee to reduce pain and improve function. Despite their potential benefits, the efficacy and biomechanical impacts of these braces require further investigation to optimize their clinical use.

Assessment of health-related quality of life (HRQoL) in patients with knee OA helps quantify disease burden and treatment effectiveness. Instruments such as the Knee Injury and Osteoarthritis Outcome Score (KOOS) and the Visual Analog Pain Scale (VAS) are commonly used to evaluate impairment and pain, respectively.

As the prevalence of knee OA continues to increase, there is a clear need for ongoing research into effective management strategies, including orthotic interventions. Understanding the impact of these approaches on quality of life and functional outcomes is essential to guide clinical decision-making.

1.2 Rationale Although several studies have examined knee braces in OA, there remains limited understanding of their specific biomechanical effects and correlation with patient-reported outcomes. The influence of braces on knee adduction moments-a key factor in medial compartment loading and pain-remains insufficiently characterized.

This study is designed to address that gap by integrating objective gait analysis with patient-reported outcomes. Assessing changes in knee adduction moments and other gait parameters will provide insight into the mechanical effectiveness of the ROAM OA Single Upright Brace. Evaluating patient-reported outcomes such as pain, comfort, and function will clarify how mechanical improvements correspond to perceived clinical benefit.

1.3 Device Description The ROAM OA knee brace, manufactured by Enovis, is intended for individuals with symptoms, physical findings, or radiographic evidence of moderate to severe unicompartmental knee OA, postoperative meniscal repair where unicompartmental unloading is indicated, or varus-valgus conditions that may benefit from compartmental unloading.

It is a single-patient-use device that alleviates pain due to single-compartment OA by applying controlled forces to the leg to shift load from the affected knee compartment to the healthier one.

1.4 Clinical Data to Date This is the first clinical study to collect prospective data on the ROAM OA knee brace.

STUDY DESIGN 2.1 Number of Study Sites Subjects will be recruited from Midwest Orthopedics at Rush and all affiliated clinical locations. All study activities will be conducted in the Rush Department of Orthopedic Surgery Motion Analysis Laboratory.

2.2 Number of Subjects Thirty subjects will be enrolled.

2.3 Estimated Study Duration Enrollment is expected at a rate of approximately two subjects per month, with clinical follow-up at four and eight weeks. The total study duration is estimated at 18 months.

STUDY OBJECTIVES 3.1 Primary Objective Biomechanical Comparison: To compare the immediate and short-term biomechanical effects of the ROAM OA brace and the Ossur Unloader One brace, focusing on knee adduction moments and spatiotemporal gait parameters.

Long-term Efficacy: To evaluate the long-term effectiveness of the ROAM OA brace in improving pain and functional outcomes among individuals with knee OA.

3.2 Secondary Objectives Evaluate safety and comfort of the ROAM OA brace, including any adverse effects and user experience.

Assess changes in gait parameters over time to determine the brace's role in promoting functional mobility and reducing medial knee load.

STUDY ENDPOINTS 4.1 Primary Endpoints Changes in Knee Adduction Moment: Measured at baseline (no brace), immediately after fitting each brace, and at four- and eight-week follow-ups using markerless gait analysis.

VAS Pain Changes: Pain levels assessed via VAS at each study milestone, including baseline, post-fitting, and follow-ups.

4.2 Secondary Endpoints Brace comfort and user compliance

Pain medication usage

KOOS score changes

Device-related and serious adverse event rate

Changes in spatiotemporal gait parameters (step length, walking speed, cadence)

STUDY POPULATION 5.1 Eligibility Criteria Inclusion Criteria

Adults aged 40-85 years

BMI <35

Diagnosed with medial compartment knee OA

Walking pain ≥4 on the VAS

Willingness to wear the assigned brace daily and complete study follow-up

Ability to walk independently for at least 20 minutes

Stable use of over-the-counter pain medications

No intra-articular injections within three months of enrollment

Exclusion Criteria

Lateral or patellofemoral OA

Previous knee joint replacement

Ligamentous instability or acute lower extremity injury

Neurological disorders affecting gait

Dermatologic or allergic conditions preventing brace use

Current use of opioids or corticosteroids

Inability to understand study instructions

Pregnancy

STUDY PROCEDURES

All participants will provide electronic informed consent through a secure platform prior to participation.

Subjects will undergo baseline data collection, brace fitting, crossover gait analysis, and randomized assignment to either brace or standard-of-care control groups. Follow-up assessments will occur at four and eight weeks, including ROM evaluation, PROMs, gait analysis, and safety review.

All data will be documented on case report forms and securely stored in accordance with institutional requirements.

Subjects will incur no cost for participation. Both braces will be provided for study purposes.

RISK/BENEFIT ASSESSMENT 7.1 Risk Category Low risk.

7.2 Potential Risks Minor risk of falls during walking tests

Temporary muscle soreness

Skin irritation from the brace

Finger strain from adjusting buckles

Emotional discomfort from questionnaires

7.3 Protection Against Risks Participants will be monitored closely, and any protocol deviations required for safety will be reported to the IRB.

7.4 Potential Benefits Participants may experience improved comfort, pain relief, or mobility due to brace use. Data collected may contribute to improved clinical management of knee OA in the future.

STATISTICAL PLAN

P-values less than 0.05 will be considered statistically significant.

8.1 Primary Analysis Changes in knee adduction moments, gait parameters, and VAS pain scores across defined timepoints will be analyzed using appropriate statistical models for repeated measures.

8.2 Secondary Analysis Secondary endpoints, including KOOS changes, brace comfort, and adverse event rates, will be analyzed descriptively and inferentially as applicable.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria:
* Age 40-85 years.
* BMI ≤ 35.
* Physician-diagnosed medial compartment knee osteoarthritis.
* Visual Analog Scale (VAS) walking pain ≥ 4.
* Willing to wear assigned brace ≥ 4 hours/day.
* Able to walk independently for 20 minutes unaided.
* Stable pain medication regimen ≥ 4 weeks.
* ≥3 months since last hyaluronic acid (HA), platelet-rich plasma (PRP), or steroid injection.

Exclusion Criteria:

* Lateral or patellofemoral osteoarthritis.
* Prior knee replacement.
* Significant ligament injury or acute lower limb injury.
* Neurological condition affecting gait.
* Severe psychiatric or neurological disorder affecting pain perception.
* Skin condition or allergy preventing brace use.
* Current use of another brace or assistive device.
* Recent opioid or corticosteroid use (<4 weeks).
* Pregnant.

Exclusion Criteria:

-

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Change in knee adduction moment during gait | Baseline, 4 weeks, and 8 weeks
  Change in peak knee adduction moment measured during gait analysis using instrumented motion capture and force platforms. Comparisons are made between baseline, 4 weeks, and 8 weeks.
Change in Visual Analog Scale (VAS) walking pain | Baseline, 4 weeks, and 8 weeks
  Change in walking pain measured by the Visual Analog Scale (VAS), in which participants rate their pain during walking along a 10-centimeter line ranging from 0 = no pain to 10 = worst imaginable pain. Lower scores indicate less pain and therefore a better outcome. Comparisons will be made between baseline, 4 weeks, and 8 weeks.

SECONDARY OUTCOMES:
Change in KOOS (Knee injury and Osteoarthritis Outcome Score) subscale scores | Baseline, 4 weeks, and 8 weeks
  Change in scores on the KOOS questionnaire, which includes five subscales: Pain, Symptoms, Activities of Daily Living, Sports/Recreation, and Quality of Life. Each subscale is scored from 0 to 100, where 0 = extreme problems and 100 = no problems. Higher scores indicate better outcomes. Comparisons will be made between baseline, 4 weeks, and 8 weeks.
Change in knee range of motion (ROM) | Baseline, 4 weeks, and 8 weeks
  Change in knee range of motion (flexion and extension) measured using goniometry; comparisons made between baseline, 4 weeks, and 8 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hochberg MC, Altman RD, April KT, Benkhalti M, Guyatt G, McGowan J, Towheed T, Welch V, Wells G, Tugwell P; American College of Rheumatology. American College of Rheumatology 2012 recommendations for the use of nonpharmacologic and pharmacologic therapies in osteoarthritis of the hand, hip, and knee. Arthritis Care Res (Hoboken). 2012 Apr;64(4):465-74. doi: 10.1002/acr.21596. PMID 22563589
- [Background] Chang J, Yuan Y, Fu M, Wang D. Health-related quality of life among patients with knee osteoarthritis in Guangzhou, China: a multicenter cross-sectional study. Health Qual Life Outcomes. 2023 May 27;21(1):50. doi: 10.1186/s12955-023-02133-x. PMID 37244981